CLINICAL TRIAL: NCT03526354
Title: A Multi-center, Randomized, Controlled Trial of Brexpiprazole for the Treatment of Co-occurring Schizophrenia and Substance Use Disorder
Brief Title: Controlled Trial of Brexpiprazole For The Treatment of Co-occurring Schizophrenia and Substance Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Massachusetts General Hospital (Other); University of North Carolina, Chapel Hill (Other); Otsuka Pharmaceutical Co., Ltd. (Industry); Augusta University (Other)
Responsible Party: Principal Investigator, Xiaoduo Fan, MD, MPH, Associate Professor of Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14611
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Substance Use Disorders
Keywords: Schizophrenia; Schizoaffective Disorder; Substance Use Disorders; Alcohol Use Disorder; Cannabis Use Disorder; Cocaine Use Disorder; Heroin Use Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Alcoholism | interventions — brexpiprazole; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Brexpiprazole 4mg daily for 12 weeks
  Interventions: Drug: Brexpiprazole
- Treatment as Usual (Active Comparator): Stay on current antipsychotic medication for 12 weeks
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole 4mg daily for 12 weeks
  Other Names: Study Medication
  Arms: Experimental
Other: Treatment as Usual — Current antipsychotic medication for 12 weeks
  Other Names: Current Antipsychotic Treatment
  Arms: Treatment as Usual

SUMMARY:
The proposed study is a 4-site, 12-week, novel, feasibility, investigation of patients who have co-occurring diagnoses of schizophrenia and current substance use disorder (alcohol, cocaine, heroin, or cannabis). Thirty-nine participants will be randomly assigned to switch to brexpiprazole (the brexpiprazole group) or remain on the same antipsychotic treatment (the control group). The study will be conducted at 4 sites in the US. The investigators expect to enroll 80 subjects across 3 sites. UMass Medical School, Worcester MA is the lead site. Sub-sites include Massachusetts General Hospital (MGH) and the University of North Carolina at Chapel Hill (UNC).

DETAILED DESCRIPTION:
STUDY OBJECTIVES

The primary objectives of the study include:

1. examine the effect of brexpiprazole treatment on the number of days of substance use in the past week as measured by the Timeline Follow-Back (TLFB) assessment;
2. examine the effect of brexpiprazole treatment on substance craving using 100-mm visual analogue scale (VAS).

The secondary objectives are to examine the effect of brexpiprazole treatment on:

1. the dollar amount spent on substances in the past week;
2. the psychiatric symptoms as measured by various clinical rating scales
3. quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Meets the DSM-5 criteria for diagnoses of schizophrenia or schizoaffective disorder and substance use disorder (alcohol, cocaine, heroin, or cannabis) based on the Mini International Neuropsychiatric Interview for the DSM-5 (MINI 7.0)
3. Uses substance on at least 4 of the past 30 days prior to randomization with at least one use in the week prior to randomization for one of substances (cocaine, heroin, cannabis or alcohol) assessed by the TLFB interview
4. Stable dose of antipsychotic agent for at least one month
5. Well established compliance with outpatient medications
6. Female subjects of child-bearing potential are required to practice appropriate birth control methods during the study.

Exclusion Criteria:

1. Psychiatrically unstable
2. Currently meets DSM-5 criteria for any substance use disorder other than caffeine, nicotine, alcohol, cocaine, heroin and cannabis
3. Significant, unstable medical conditions including severe cardiovascular, hepatic, renal or other medical diseases
4. History of a seizure disorder
5. Pregnancy or breastfeeding
6. Currently on aripiprazole or cariprazine
7. Currently on medications to treat substance use (disulfiram, naltrexone, acamprosate, methadone, buprenorphine, varenicline or buproprion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (4):
- United States (4):
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan X, Freudenreich O, Jarskog LF, McEvoy J, Harrington A. Brexpiprazole for the Treatment of Co-occurring Schizophrenia and Substance Use Disorder: A Multisite, Randomized, Controlled Trial. J Clin Psychiatry. 2025 Oct 13;86(4):25m15786. doi: 10.4088/JCP.25m15786. PMID 41129678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Treatment as Usual
Started | 21 | 18
Completed | 15 | 14
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Treatment as Usual | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (12.0) | 39.8 (11.2) | 37.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 16 | 14 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 9 | 17
  African American | 9 | 10 | 19
  Other | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Timeline Follow Back (TLFB)
Description: The Timeline Follow Back (TLFB) scale is used to measure weekly substance use for alcohol, marijuana, cocaine, and/or heroin by assessing the number of days a person used substances in the past week, on a scale from 0 to 7 [0 = no substances that week; 7 = substance use every day]. The outcome measure was the number of days per week that participants used a substance. If participants use more than one substance, only the primary substance (one used mostly frequently) was analyzed.
  While the TLFB was assessed weekly, the outcome measure reported is the change in substance use between Week 0 (Baseline) and Week 12 (End of Study). A decrease in number of days/week that substances were used indicates an improved (better) outcome.
  While the TLFB was assessed weekly, the outcome measure reported is the change in substance use between Week 0 (Baseline) and Week 12 (End of Study). A decrease in number of days/week that substances were used indicates an improved (better) outcome.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
score on a scale | -1.765 [-3.117 to -.413] | -.532 [-1.910 to .846]

2. Primary Outcome: Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) measures substance craving. Subjects will make a mark on an unlabeled 100-millimeter line indicating their desire to use a particular substance over the past 7-days. A score of 0 indicates no desire to use and 100 indicating the strongest desire to use possible. The assessment was done weekly. Subjects reported craving for any substances they used that week with a separate mark for each substance (e.g., a mark for alcohol craving and another mark for marijuana). For outcome measures, only the primary substance (the substance used most frequently, as determined by the Timeline Follow Back assessment) was included. While cravings were assessed weekly, only the change in craving from Week 0 (Baseline) to Week 12 (End of Study) is reported; a decreased score (reduction in cravings) represents an improved outcome.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
score on a scale | -33.421 [-49.305 to -17.536] | -8.898 [-25.511 to 7.716]

3. Secondary Outcome: Amount of Money Spent on Substances
Description: The amount of money spent on substances over a 7-day period will also be recorded as part of each weekly visit. Decreased money spent on substances over a 7-day period will also be considered an improved outcome.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: dollars spent
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
dollars spent | -20.974 [-51.647 to 9.700] | 14.605 [-16.497 to 45.707]

4. Secondary Outcome: Positive and Negative Symptom Scale (PANSS)
Description: The Positive and Negative Symptom Scale (PANSS) is a measure used to assess symptom severity in patients with schizophrenia. Each item (symptom) is scored on a 7-point scale (1 = absent and 7 = extreme). The minimum and maximum values for the total 30 items (PANSS Total Score) are 30 and 210 respectively. Higher scores represent higher levels of psychiatric symptoms (worse outcomes).
  The PANSS has three subscales: "Positive" (measuring positive symptoms), "Negative" (measuring negative symptoms), and "General Psychopathology" (measuring general psychiatric symptoms). There are 7 items each for Positive and Negative subscales (minimum value for each is 7, and maximum value is 49), and 16 items for General Psychopathology (minimum value is 16 and maximum is 112).
  This study looked at changes in all 3 subscales and the PANSS total score between Week 0 (Baseline) and Week 12 (End of Study), with a decrease in score indicating improved psychiatric functioning.
Time Frame: 12 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
score on a scale | -3.690 [-9.188 to 1.807] | -.274 [-5.996 to 5.447]

5. Secondary Outcome: Clinical Global Impression - Severity
Description: The Clinical Global Impression - Severity (CGI-S) measures illness severity on a 7-point Likert scale, with a higher score indicating higher illness severity and worse outcomes (1 = "Normal, not at all ill" and 7 = "Among the most extremely ill patients"). The outcome measure for this study looked at the change in the CGI-S score between Week 0 (Baseline) and Week 12 (end of study), with a reduction in score indicating improved outcomes.
Time Frame: 12 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
score on a scale | -.320 [-.601 to -.038] | -.128 [-.413 to .156]

6. Secondary Outcome: Heinrichs Carpenter Quality of Life Scale (QOL)
Description: The Heinrichs Carpenter Quality of Life Scale (QOL)is a 21-item scale providing information on symptoms and functioning in patients with schizophrenia. Items are scored on a 0-6 scale, with 0 being no evidence of that item (e.g., social relationships are virtually absent) and 6 being adequate evidence of that item (e.g., adequate social relationships). Two items (#1 - "Intimate relationship with household members" and # 12 - "Satisfaction with occupational role functioning") are scored a "9" if the item is not applicable (e.g., lives alone with no close family or does not have an occupational role). Therefore, total scores can range from 0 to 132 (if 9s are scored). A higher total score indicates better psychosocial functioning.
  For this study, the outcome measure looked at the change in total score between Week 0 and Week 12.
Time Frame: 12 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental | Treatment as Usual
Number analyzed (Participants) | 21 | 18
score on a scale | 4.049 [-1.950 to 10.049] | -5.146 [-11.293 to 1.001]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant's screening through their study completion (Week 12 or Early Termination), an average of 3 months.
Arm/Group | Experimental | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 10/21 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=21) | Treatment as Usual (N=18)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigure/Tiredness (General disorders) | 3 (3) | 0 (0)
Dizziness (General disorders) | 2 (2) | 1 (1)
Cold-like symptoms (General disorders) | 2 (2) | 3 (3)
Trouble Sleeping (General disorders) | 2 (2) | 0 (0)
Nausea (General disorders) | 3 (3) | 2 (2)
Restlessness/Irritability (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT03526354/Prot_SAP_000.pdf